CLINICAL TRIAL: NCT05447351
Title: Effects of Personalized Dietary and Lifestyle Treatments on the Reduction of Cardiovascular and Metabolic Risk in Overweight and Obese Patients
Brief Title: Beneficial Effects of Dietary and Lifestyle Change in Overweight and Obese Subjects
Acronym: Healthy-MET
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, piero portincasa, Professor, MD, University of Bari
Other Study IDs: HEALTHYMET01-2022
Record Dates: First submitted 2022-06-22; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Overweight and Obesity; Cardiovascular Diseases; Metabolic Syndrome; Non-Alcoholic Fatty Liver Disease
Keywords: Overweight and Obesity; Cardiovascular diseases; Mediterranean Diet; Lifestyle; Physical activity; Metabolic disorders
MeSH Terms: conditions — Overweight; Obesity; Cardiovascular Diseases; Metabolic Syndrome; Non-alcoholic Fatty Liver Disease; Motor Activity; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — * bio-humoral indicators of metabolic homeostasis (glyco-lipid profile, adipokines, insulinemia, HOMA index) and pro-inflammatory status (serum interleukins, amyloid A, CRP)
  * bio-humoral dosage of hormones involved in the metabolism of intestinal nutrients (GLP-1, GIP, total and acylated ghrelin, PYY)
  * profiling of gut microbiota and assessment of metabolome
  * ultrasonographic measurement of fatty liver and visceral fat accumulation
  * marker of intestinal permeability (blood / urine dosage of LPS, zonulin)
  * urinary dosage of sugars with selective gastrointestinal absorption, aimed at evaluating intestinal permeability at the gastric, ileal and colic level
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treated: Counselling, personalized dietary strategy aimed at increasing the adherence to Mediterranean diet, personalized physical activity program with a personal trainer, use of digital tools (i.e., games, apps) aimed at improving the adherence to dietary/lifestyle indications.
- Control: generic dietary indications oriented to weight reduction; generic invitations to increase physical activity, routine monitoring

SUMMARY:
Obesity and overweight are noncommunicable diseases with increasing incidence in children, adolescents and adults. In 2016, more than 1.9 billion adults aged 18 and over were overweight and over 650 million were obese (WHO). In the EU-27 (Eurostat data), 45.7% of women and 60.2% of men were overweight, while 16.3% and 16.8%, respectively, were obese. The growing incidence of overweight and obesity generate worldwide increasing incidence of related conditions as cardiovascular diseases, diabetes, metabolic disorders, and cancer, with relevant socio-economical (increase in health costs, increase in disabilities) and environmental consequences (unsustainability of food models, increase in ecological footprint, worsening of climate changes). A transformation of food systems and individual behaviours are necessary to improve the quality of life and the sustainability of lifestyle, which should be oriented at preventing o treating overweight and obesity.

DETAILED DESCRIPTION:
The study is aimed to measure the beneficial effects of specific dietary models (i.e., Mediterranean Diet) and healthy lifestyle (i.e., controlled physical activity) in reducing body/organ fat accumulation and in the improvement of metabolic health. A comprehensive and combined analysis of these effects (mainly following personalized strategies and close follow-up) on pathogenic mechanisms affecting cardiovascular and metabolic risk, pro-inflammatory status and intestinal permeability in the medium-long term is still lacking.

During the study, overweight/obese subjects (i.e. Body Mass Index equal or higher to 25Kg/m2) will be assessed at basal and monitored during a 24 months follow-up

ELIGIBILITY:
Inclusion Criteria:

* overweight or obese patients
* patients who able to sign informed consent

Exclusion Criteria:

* failure to sign informed consent;
* inclusion in other research protocols
* Normal weight patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Enrolled in the study will be 200 overweight or obese adult patients (comparable sex ratio) entering the outpatient clinic for metabolic diseases.
  Subjects will be randomized in two groups (i.e., n=100 treated and n=100 controls). For an unpaired t-test (i.e., comparison of two groups), 50 is the minimum sample size needed in each group to obtain a power of 0.80, when the effect size is medium and a significance level of 0.05 is employed.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Effects of treatments on Body Mass Index and waist circumference | 24 months
  waist circumference will be measured and expressed in cm. weight and height will be combined to report BMI in kg/m^2. Measurements will be taken at enrollment and during follow-up.
Effects of treatments on visceral fat | 24 months
  Measurement of visceral fat by ultrasonography (expressed in mm) will be performed at baseline and during follow-up

SECONDARY OUTCOMES:
Change in metabolic indices and in hormones involved in the regulation of glucose metabolism | 24 months
  gluco-lipid profile, adipokines, insulinemia, HOMA index will be measured at baseline and during the follow-up
Change in hormones involved in nutrient sensing | 24 months
  GLP-1, GIP, total and acylated ghrelin, PYY will be measured at baseline and during the follow-up
Effects of microbiota and metabolome | 24 months
  profiling of gut microbiota and assessment of metabolome will be assessed in enrolled subjects at baseline and during follow-up
Effects on intestinal permeability | 24 months
  markers of intestinal permeability (blood / urine dosage of LPS, zonulin) urinary dosage of sugars with selective gastrointestinal absorption, aimed at evaluating intestinal permeability at the gastric, ileal and colic level. Assessments will be performed at baseline and during the follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Biomedical Sciences and Human Oncology - Clinica medica "A. Murri", Bari, BA, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yarnoz-Esquiroz P, Olazaran L, Aguas-Ayesa M, Perdomo CM, Garcia-Goni M, Silva C, Fernandez-Formoso JA, Escalada J, Montecucco F, Portincasa P, Fruhbeck G. 'Obesities': Position statement on a complex disease entity with multifaceted drivers. Eur J Clin Invest. 2022 Jul;52(7):e13811. doi: 10.1111/eci.13811. Epub 2022 May 12. PMID 35514242
- [Background] Portincasa P, Bonfrate L, Khalil M, Angelis M, Calabrese FM, D'Amato M, Wang DQ, Di Ciaula A. Intestinal Barrier and Permeability in Health, Obesity and NAFLD. Biomedicines. 2021 Dec 31;10(1):83. doi: 10.3390/biomedicines10010083. PMID 35052763
- [Background] Di Ciaula A, Bonfrate L, Krawczyk M, Fruhbeck G, Portincasa P. Synergistic and Detrimental Effects of Alcohol Intake on Progression of Liver Steatosis. Int J Mol Sci. 2022 Feb 27;23(5):2636. doi: 10.3390/ijms23052636. PMID 35269779
- [Background] Baldini F, Khalil M, Serale N, Voci A, Portincasa P, Vergani L. Extent and features of liver steatosis in vitro pave the way to endothelial dysfunction without physical cell-to-cell contact. Nutr Metab Cardiovasc Dis. 2021 Nov 29;31(12):3522-3532. doi: 10.1016/j.numecd.2021.08.032. Epub 2021 Aug 13. PMID 34629256
- [Background] Vecchie A, Dallegri F, Carbone F, Bonaventura A, Liberale L, Portincasa P, Fruhbeck G, Montecucco F. Obesity phenotypes and their paradoxical association with cardiovascular diseases. Eur J Intern Med. 2018 Feb;48:6-17. doi: 10.1016/j.ejim.2017.10.020. PMID 29100895
- [Background] Bonfrate L, Wang DQ, Garruti G, Portincasa P. Obesity and the risk and prognosis of gallstone disease and pancreatitis. Best Pract Res Clin Gastroenterol. 2014 Aug;28(4):623-35. doi: 10.1016/j.bpg.2014.07.013. Epub 2014 Jul 22. PMID 25194180
- [Background] Faienza MF, Wang DQ, Fruhbeck G, Garruti G, Portincasa P. The dangerous link between childhood and adulthood predictors of obesity and metabolic syndrome. Intern Emerg Med. 2016 Mar;11(2):175-82. doi: 10.1007/s11739-015-1382-6. Epub 2016 Jan 12. PMID 26758061
- [Background] Di Ciaula A, Portincasa P. Diet and Contaminants: Driving the Rise to Obesity Epidemics? Curr Med Chem. 2019;26(19):3471-3482. doi: 10.2174/0929867324666170518095736. PMID 28521687
- [Background] Faienza MF, Chiarito M, Molina-Molina E, Shanmugam H, Lammert F, Krawczyk M, D'Amato G, Portincasa P. Childhood obesity, cardiovascular and liver health: a growing epidemic with age. World J Pediatr. 2020 Oct;16(5):438-445. doi: 10.1007/s12519-020-00341-9. Epub 2020 Feb 4. PMID 32020441
- [Background] Baldini F, Khalil M, Bartolozzi A, Vassalli M, Di Ciaula A, Portincasa P, Vergani L. Relationship between Liver Stiffness and Steatosis in Obesity Conditions: In Vivo and In Vitro Studies. Biomolecules. 2022 May 23;12(5):733. doi: 10.3390/biom12050733. PMID 35625660
- [Background] Di Palo DM, Garruti G, Di Ciaula A, Molina-Molina E, Shanmugam H, De Angelis M, Portincasa P. Increased Colonic Permeability and Lifestyles as Contributing Factors to Obesity and Liver Steatosis. Nutrients. 2020 Feb 21;12(2):564. doi: 10.3390/nu12020564. PMID 32098159
- [Background] Bonfrate L, Di Palo DM, Celano G, Albert A, Vitellio P, De Angelis M, Gobbetti M, Portincasa P. Effects of Bifidobacterium longum BB536 and Lactobacillus rhamnosus HN001 in IBS patients. Eur J Clin Invest. 2020 Mar;50(3):e13201. doi: 10.1111/eci.13201. Epub 2020 Feb 12. PMID 31960952
- [Background] Vacca M, Celano G, Calabrese FM, Portincasa P, Gobbetti M, De Angelis M. The Controversial Role of Human Gut Lachnospiraceae. Microorganisms. 2020 Apr 15;8(4):573. doi: 10.3390/microorganisms8040573. PMID 32326636
- [Background] Di Ciaula A, Baj J, Garruti G, Celano G, De Angelis M, Wang HH, Di Palo DM, Bonfrate L, Wang DQ, Portincasa P. Liver Steatosis, Gut-Liver Axis, Microbiome and Environmental Factors. A Never-Ending Bidirectional Cross-Talk. J Clin Med. 2020 Aug 14;9(8):2648. doi: 10.3390/jcm9082648. PMID 32823983
- [Background] Vitellio P, Celano G, Bonfrate L, Gobbetti M, Portincasa P, De Angelis M. Effects of Bifidobacterium longum and Lactobacillus rhamnosus on Gut Microbiota in Patients with Lactose Intolerance and Persisting Functional Gastrointestinal Symptoms: A Randomised, Double-Blind, Cross-Over Study. Nutrients. 2019 Apr 19;11(4):886. doi: 10.3390/nu11040886. PMID 31010241
- [Background] Molina-Molina E, Shanmugam H, Di Ciaula A, Grattagliano I, Di Palo DM, Palmieri VO, Portincasa P. (13C)-Methacetin breath test provides evidence of subclinical liver dysfunction linked to fat storage but not lifestyle. JHEP Rep. 2020 Nov 4;3(1):100203. doi: 10.1016/j.jhepr.2020.100203. eCollection 2021 Feb. PMID 33490935
- [Background] Cosola C, Rocchetti MT, di Bari I, Acquaviva PM, Maranzano V, Corciulo S, Di Ciaula A, Di Palo DM, La Forgia FM, Fontana S, De Angelis M, Portincasa P, Gesualdo L. An Innovative Synbiotic Formulation Decreases Free Serum Indoxyl Sulfate, Small Intestine Permeability and Ameliorates Gastrointestinal Symptoms in a Randomized Pilot Trial in Stage IIIb-IV CKD Patients. Toxins (Basel). 2021 May 5;13(5):334. doi: 10.3390/toxins13050334. PMID 34063068
- [Background] Rizzello CG, Portincasa P, Montemurro M, Di Palo DM, Lorusso MP, De Angelis M, Bonfrate L, Genot B, Gobbetti M. Sourdough Fermented Breads are More Digestible than Those Started with Baker's Yeast Alone: An In Vivo Challenge Dissecting Distinct Gastrointestinal Responses. Nutrients. 2019 Dec 4;11(12):2954. doi: 10.3390/nu11122954. PMID 31817104
- [Background] Van Gorp H, Huang L, Saavedra P, Vuylsteke M, Asaoka T, Prencipe G, Insalaco A, Ogunjimi B, Jeyaratnam J, Cataldo I, Jacques P, Vermaelen K, Dullaers M, Joos R, Sabato V, Stella A, Frenkel J, De Benedetti F, Dehoorne J, Haerynck F, Calamita G, Portincasa P, Lamkanfi M. Blood-based test for diagnosis and functional subtyping of familial Mediterranean fever. Ann Rheum Dis. 2020 Jul;79(7):960-968. doi: 10.1136/annrheumdis-2019-216701. Epub 2020 Apr 20. PMID 32312770
- [Background] Portincasa P, Bonfrate L, Vacca M, De Angelis M, Farella I, Lanza E, Khalil M, Wang DQ, Sperandio M, Di Ciaula A. Gut Microbiota and Short Chain Fatty Acids: Implications in Glucose Homeostasis. Int J Mol Sci. 2022 Jan 20;23(3):1105. doi: 10.3390/ijms23031105. PMID 35163038